CLINICAL TRIAL: NCT06329284
Title: Midkine Interplays With Oxidative Stress and Inflammatory Milieu to Induce Preeclampsia in Normotensive Pregnant Women
Brief Title: Midkine Role With Deregulated Oxidative and Immune Milieu in Induction of Preeclampsia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Shereen Naguib, Lecturer of Obstetrics & Gynecology, Faculty of Medicine, Benha University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RC 31.1.2024
Record Dates: First submitted 2024-03-10; First posted 2024-03-25 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Pre-Eclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Intervention Model Description: Newly pregnant normotensive (NT) women with singleton fetus
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Serum Midkine (Other)
  Interventions: Diagnostic Test: ELISA

INTERVENTIONS:
Diagnostic Test: ELISA — ELISA estimation of serum Midkine, tumor necrosis factor Alfa, superoxide dismutase, malondialdehyde, placental growth factor and placental soluble fms-like tyrosine kinase 1

SUMMARY:
Preeclampsia (PE) is a hypertensive pregnancy-related disorder that endangers maternal and fetal outcomes and accounts for 9-10% of maternal mortalities with its early-onset phenotype is the most dangerous, but its etiology is still not fully elucidated.

Midkine (MDK) is a multifunctional protein that plays a unique role in the development of hypertension (HTN), via its proatherogenic effect and induction of overexpression of angiotensin converting enzyme. Oxidative stress (OS) upregulates the expression of MDK and MDK induces propagation of neoangiogenesis and acts as chemotactic for neutrophils.

ELIGIBILITY:
Inclusion Criteria:

* Newly pregnant normotensive (NT) women with singleton fetus;
* Free of the Exclusion Criteria.

Exclusion Criteria:

* Women with history of complicated pregnancy;
* Had manifest essential hypertension, Diabetes Mellitus or chronic kidney diseases;
* Had multiple gestational sacs, morbid obesity with Body Mass Index at time of pregnancy diagnosis over 35 kg/m2;
* Had genetic disorders, coagulopathy, autoimmune diseases or maintained on immunosuppressive therapy.

Ages: 21 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Severity of Pre-Eclampsia (PE) | 8 months
  Correlation between Serum midkine levels and blood pressure measurements

CONTACTS AND LOCATIONS:
Locations (1):
- Banha University, Banhā, El- Qalyobia, Egypt